CLINICAL TRIAL: NCT00767715
Title: A Randomized Open Label Study on the Efficacy, Tolerability, and Total Costs of Olanzapine Versus Conventional Antipsychotics in the Treatment of Acute Mania in Sweden
Brief Title: A Study in the Treatment of Acute Mania
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Trial discontinued due to low enrollment
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7313; F1D-SO-HGLY
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Last update posted 2008-10-07 (Estimated); Status verified 2008-10

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Olanzapine; Haloperidol; Clopenthixol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Patients will be given olanzapine
  Interventions: Drug: olanzapine
- B (Active Comparator): Patients will be given either haloperidol or zuclopentixol
  Interventions: Drug: haloperidol; Drug: zuclopentixol

INTERVENTIONS:
Drug: olanzapine — physician determined dose, oral, daily, 5 months
  Other Names: LY170053; Zyprexa
  Arms: A
Drug: haloperidol — physician determined dose, oral, parenteral (<= 3 days), daily, 5 months
  Arms: B
Drug: zuclopentixol — physician determined dose, oral, parenteral (<= 3 days), daily, 5 months
  Arms: B

SUMMARY:
The purpose of this study is to test the efficacy and total costs of olanzapine versus commonly used conventional antipsychotics in Sweden.

DETAILED DESCRIPTION:
The primary objective is to show that the efficacy of olanzapine is non-inferior to the conventional antipsychotics haloperidol or zuclopentixol in the treatment of an acute manic or mixed episode of bipolar disorder. Efficacy is defined as time to remission, as measured by the total scores of the Young Mania Rating Scale (Y-MRS), MADRS-S, and Clinical Global Impression - Bipolar (CGI-BP). Time from baseline to remission is defined as the primary efficacy measure. Remission is defined as a Y-MRS score <=12 AND a MADRS-S score <=12 AND CGI-BP = 1 or 2.

Secondary efficacy assessments will include time from baseline to

* Response, as defined as a reduction of Y-MRS score greater than or equal to 50% compared to baseline
* Relapse of mania, as defined as a Y-MRS score >= 16 AND CGI-BP >2 after having met the criteria for remission
* Switch into depression, as defined as a MADRS-S score >=17 AND fulfilled criteria for Major Depression as self-assessed by DSRS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar I disorder and currently display an acute manic or mixed episode (with or without psychotic features)
* Patients must have a Y-MRS total score of greater or equal to 20 at visit 2
* Patients must have experienced at least one manic or mixed episode prior to study enrollment
* Female of childbearing potential must be using a medically accepted means of contraception, or practice sexual abstinence
* Each patient must have a level of understanding sufficient to communicate intelligently with study personnel
* Patients must be considered reliable
* Each patient must understand the nature of the study and signed informed consent

Exclusion Criteria:

* Female patients who are pregnant or lactating
* Serious, unstable illnesses such that hospitalization for the disease is anticipated within 3 month or death is anticipated within 3 years
* Uncorrected hypothyroidism or hyperthyroidism
* Narrow-angle glaucoma
* History of allergic reactions or intolerance to study medications
* DSM-IV substance dependence within the past 30 days at the judgement of the investigator
* Judged clinically to be at serious suicidal risk
* Treatment with an injectable depot neuroleptic within less than one dosing interval between depot neuroleptic injections prior to visit 2
* Any patient treated with clozapine within 4 weeks prior to visit 2
* Subjects who have received treatment with ECT within one month prior to visit 1

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2004-10; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Time to remission by Young Mania Rating Scale, MADRS-S and CGI-BP | 5 months

SECONDARY OUTCOMES:
Resource utilization Clinical Report Form (RUCRF) | 5 months
Disability free day assessment (DFDA) | 5 months
Medication compliance | 5 months
Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) | 5 months
Euro Qol instrument | 5 months
Drug Attitude Inventory (DAI) | 5 months
Response by Y-MRS | 5 months
Frequency of and time to relapse into mania by Y-MRS and CGI-BP | 5 months
Frequency of and time to switch to depression by MADRS-S and DSRS | 5 months
Time to remission in patients with psychotic features by SCID-I judgement, Y-MRS item 8 and PANSS positive items mean sum | 5 months
Adverse events | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danderyd, Sweden